CLINICAL TRIAL: NCT06297993
Title: A Global Multi-Center Prospective Observational Cohort to Support Drug Development in Adult Patients With Primary Sclerosing Cholangitis (WIND-PSC)
Brief Title: Global Prospective, Observational Cohort of Adult Patients With Primary Sclerosing Cholangitis (WIND-PSC Study)
Acronym: WIND-PSC
Status: Recruiting | Type: Observational
Sponsor: PSC Partners Seeking a Cure (Other)
Responsible Party: Sponsor
Other Study IDs: WIND-PSC-01
Record Dates: First submitted 2024-01-29; First posted 2024-03-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: PSC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A standardized procedure for collection and processing of human blood will be applied to all blood samples collected as part of the study. Barcoded samples will be stored at the clinical centers, and corresponding data will be entered into the study database. Any protocol deviations should also be recorded by each center.
  30mL of blood is collected at baseline and at each annual visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with a confirmed diagnosis of large duct PSC.: 1. Adult patients between 18 and 75 years of age (inclusive) who can comprehend instructions, follow the study procedures and are willing to sign an Informed Consent Form (ICF).
  2. Confirmed clinical diagnosis of large duct PSC

SUMMARY:
Develop an appropriate real-world data comparator cohort to support the design, execution, and serve as an external control for interventional clinical trials in PSC.

DETAILED DESCRIPTION:
Global, multi-center longitudinal observational cohort study. Collection of prospective clinical data to include liver-related clinical outcomes and safety events, hepatobiliary malignancies, relevant key biomarkers, imaging assessments, PSC-related clinical symptoms, patient-reported outcomes, and medication use in adult patients with PSC.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between 18 and 75 years of age (inclusive) who can comprehend instructions, follow the study procedures and are willing to sign an Informed Consent Form (ICF).
2. Confirmed clinical diagnosis of large duct PSC.

Exclusion Criteria:

1. Clinically significant acute or chronic liver disease of an etiology other than PSC (including but not limited to metabolic-dysfunction associated steatohepatitis (MASH), PBC, HCV, HBV, or alcoholic hepatitis, Wilson's disease, alpha-1 antitryp-sin deficiency, acute or chronic drug-induced liver injury)

   * Patients with PSC and elements of AIH overlap are allowed to enroll
   * Patients with metabolic dysfunction associated steatotic liver disease (MASLD) or benign steatosis are allowed to enroll
2. Small-Duct PSC.
3. Clinically diagnosed secondary or IgG4-related sclerosing cholangitis.
4. Clinically diagnosed infections (including acute cholangitis) and receiving treatment within the past 7 days; patients on chronic suppressive antibiotics for acute cholangitis will be allowed to enroll
5. Hospitalization in the past 7 days
6. UDCA dose >28 mg/kg
7. Evidence of current or historical decompensated cirrhosis based on the following clinical events:

   * Ascites > Grade 2 and requiring treatment
   * Esophageal or gastric variceal bleeding requiring hospitalization
   * Hepatic encephalopathy (as defined by a West Haven score ≥ 2)
   * Spontaneous bacterial peritonitis defined as ascites absolute neutrophil count >250/mm3 in the absence of an intra-abdominal source of infection
   * AKI-HRS according to AASLD Guidelines (Flamm 2021)
   * Portal hypertension based on a platelet count < 150 × 109/L and LSM > 15 kPa with clinical, laboratory, imaging and/or other relevant parameters
8. Prior liver transplantation
9. MELD 3.0 Score >15. For subjects on anticoagulation medication, baseline INR determination for MELD score calculation should take this use into account.
10. History, evidence, or high suspicion of hepatobiliary malignancies or active colon cancer based on imaging, screening laboratory values, and/or clinical symptoms. Patients with a history of colon cancer who have undergone a colectomy and have no current evidence of colon cancer will be allowed to enroll in the study.
11. Participants with current clinical or laboratory evidence of any severe, progressive, or uncontrolled disease, related or unrelated to PSC and which, in the opinion of the investigator, has an expected survival of less than 52 weeks.
12. Participants who are impaired, incapacitated, or incapable of completing study-related assessments or giving informed consent.
13. Prisoners or participants who are involuntarily incarcerated.
14. Participants who are currently participating in an investigational PSC therapy clinical study or who have participated in such a study within the past 12 weeks
15. Absence of data in medical records to assess inclusion and exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2000 adult participants with confirmed diagnosis of large duct PSC
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Develop an appropriate real-world data (RWD) comparator cohort to support the design, execution, and serve as an external control for interventional clinical trials in PSC. | Quarterly for five years from enrollment
  Collection of liver-related data including PSC symptoms, medical history, adverse events, and outcomes at enrollment and each quarterly and annual visit.

SECONDARY OUTCOMES:
Develop a large clinical and biomarker data set to identify individual and/or composite surrogate end-points likely to predict clinical benefit for use in the design of interventional studies in PSC. | Quarterly for five years from enrollment
  Collection of biomarkers at enrollment and each annual visit.
Develop a large clinical and biomarker data set to identify individual and/or composite surrogate end-points likely to predict clinical benefit for use in the design of interventional studies in PSC. | Quarterly for five years from enrollment
  Collection of imaging at enrollment and each annual visit.
Evaluate direct participant experiences with standardized tools to determine changes over time, the association with clinical events, biomarkers, and disease progression | Quarterly for five years from enrollment
  Patient Reported Outcomes surveys will be collected from all participants at enrollment and each quarterly and annual visit.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Levy, MD, Principal Investigator — University of Miami; Stephen Rossi, PharmD, Principal Investigator — PSC Partners Seeking a Cure
Locations (15):
- United States (10):
  - UC Davis, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Schiff Center for Liver Diseases / University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University Health Network, Toronto, Ontario
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany
- University of Milano Bicocca, Milan, Monza (MB), Italy
- Auckland University, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided